CLINICAL TRIAL: NCT03980379
Title: A Study of Pharmacokinetics, Efficacy, and Safety of 304 Injection Compared With Rituximab in B Cell Non-Hodgkin's Lymphoma
Brief Title: Pharmacokinetics, Efficacy and Safety of the 304 Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-304-NHL-I-02
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-05

CONDITIONS: CD20 Positive B Cell NHL
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 304 injection.WILL be administered single dose IV in the patients with CD20 positive B cell NHL
  Interventions: Drug: 304 injection
- control group (Active Comparator): Rituximab will be administered single dose IV in the patients with CD20 positive B cell NHL.
  Interventions: Drug: rituximab injection

INTERVENTIONS:
Drug: 304 injection — Monoclonal antibodies, 100mg/10ml per injection
  Arms: experimental group
Drug: rituximab injection — 100mg/10ml per injection ，manufactured by Roche
  Arms: control group

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic of the experimental drug 304 injection compared with rituximab injection in patients with CD20 positive B-cell non-Hodgkin lymphoma who had previously achieved CR/CRu status but had not deteriorated or relapsed. While to assess the safety and efficacy of the experimental drug 304 injection compared with rituximab injection.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel controlled, single-dose study to evaluate the pharmacokinetic, safety and efficacy of 304 injection compared with rituximab injection. To avoid the impact of tumor burden on pharmacokinetics, this study will be conducted in CD20 positive B-cell non-Hodgkin lymphoma patients who have achieved CR/CRu status and have not yet deteriorated or relapsed. All patients will be randomly averagely entered into the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Histological examination confirmed CD20-positive B-cell non-Hodgkin's lymphoma patients (according to WHO 2008 lymphoid tissue tumor type, and a corresponding medical history basis);
* Previous treatments with CR/CRu (see Appendix 1 for lymphoma efficacy criteria) and those with CD20-positive B-cell non-Hodgkin's lymphoma who have not yet worsened and relapsed believe that they can benefit from anti-CD20 monoclonal antibody therapy. The diagnosis of CRu requires complete raw data (using CT findings. The preferred enhanced CT examination)
* At the time of enrollment, the Eastern Oncology Cooperative Group (ECOG) had a physical status score of ≤1 (see Appendix 2 for the evaluation criteria for the ECOG physical status score) and the expected survival period was more than four months
* In the screening test, WBC≥3×109/L, HGB≥80g/L, ANC≥1.5×109/L, PLT≥75×109/L, left ventricular ejection fraction (LVEF) ) ≥ 50%
* Female patients of childbearing age were negative for the blood pregnancy test during the screening period. Patients of childbearing age are willing to contraception after signing the informed consent form until 6 months after the end of the study treatment, including but not limited to: hormonal contraception, or physical contraception, or abstinence
* Be able to understand and comply with clinical trial protocol requirements and voluntarily sign written informed consent

Exclusion Criteria:

* In the past 5 years, there have been other medical history of malignant tumors (except for local malignant tumors that have been cured, such as cutaneous basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or breast carcinoma in situ)
* Those who have used chemotherapy drugs within 4 weeks before enrollment
* The clinical half-life of more than 5 drugs after taking other clinical trials in three months or other clinical trials (whichever is longer)
* The last time you used rituximab or other anti-CD20 mAbs for no more than 4 months
* In the screening test, the liver and kidney function tests have any of the following abnormalities: total bilirubin > 1.5 times the upper limit of normal, ALT > 2.5 times the upper limit of normal, AST > 2.5 times the upper limit of normal, ALP > 2.5 times the upper limit of normal, Blood Cr>1.5 times the upper limit of normal value
* Hyperthyroidism
* He was transfused within 2 weeks before enrollment, or hematopoietic cytokine therapy, such as granulocyte colony-stimulating factor (G-CSF), thrombopoietin, erythropoietin, etc.
* Those who were vaccinated or planned to vaccinate (attenuate) live virus vaccine within 4 weeks prior to enrollment;
* Oversized surgery (not including diagnostic surgery) in the past 8 weeks;
* Have evidence or history of central nervous system involvement or cranial neuropathy;
* Treponema pallidum antibody positive, or HIV antibody positive, or HCV antibody positive;
* HBV examination showed one of the following results: a, HBsAg positive; b, although HBsAg negative, but anti-HBc positive and peripheral blood HBV DNA titer can be measured;
* Have had herpes zoster and have sequelae or latent infections;
* Patients with a history of severe heart disease, including but not limited to: New York Heart Association NYHA class II-IV heart failure (see Appendix 3 for NYHA heart failure grading), uncontrolled angina or arrhythmia, heart conduction above II Blocking, myocardial infarction occurred within 6 months
* Serious illnesses that have been or are currently suffering from any other organ or system (including but not limited to: severely active infections, uncontrolled diabetes, uncontrolled hypertension/hypotension, cerebrovascular disease, gastric ulcers, respiratory diseases, activities) Sexual autoimmune diseases, etc.; and any other medical history that the subject judges to be unsuitable for participating in the trial;
* Pregnant or lactating female subjects, or those who are unwilling to contraception during the trial
* Severe allergies, or any component known to be rituximab or other anti-CD20 mAbs or allergic to murine proteins;
* Subjects had a history of drug abuse or a history of smoking and drinking during the first 6 months of enrollment;
* The investigator judged that the patient was not suitable for entering any other circumstances of the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
AUC [0-t] | For 85 days
  To assess PK parameter of plasma 304 or rituximab: Area under the concentration-time curve from time zero to last time of quantifiable concentration (AUC [0-t])
AUC [0-∞] | For 85 days
  To assess PK parameter of plasma 304 or rituximab:
  Area under the concentration-time curve from time zero extrapolated to infinity (AUC [0-∞])
Cmax | For 85 days
  To assess PK parameter of plasma 304 or rituximab：Observed maximum plasma concentration (Cmax)

SECONDARY OUTCOMES:
tmax | For 85 days
  To assess PK parameter of plasma 304 or rituximab：Time to Cmax (tmax)
t1/2 | For 85 days
  To assess PK parameter of plasma 304 or rituximab：Elimination half-life (t1/2)
MRT | For 85 days
  To assess PK parameter of plasma 304 or rituximab：Mean residence time (MRT)
Vz | For 85 days
  To assess PK parameter of plasma 304 or rituximab：Apparent volume of distribution(Vz)
CLz | For 85 days
  To assess PK parameter of plasma 304 or rituximab：apparent clearance (CLz)
ADA | Up to 9 months
  To evaluate the incidence of anti-304 and anti-rituximab antibodies
Adverse events | Up to 85 days
  To evaluate the adverse events (incidence, severity, outcome, causality with the investigational drug, etc.).

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The 307 Hospital of People's Liberation Army, Beijing, Beijing Municipality
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Hospital of Hebei University, Baoding, Heibei
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - The First Affiliated Hospita of Zhengzhou University, Zhengzhou, Henan
  - Weihai Municipal Hospital, Weihai, Shandong
  - Tianjin Medical University Cancer Institute &Hospital, Tianjing, Tianjing
  - The Second Affiliated Hospital of Soochow University, Suzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided